CLINICAL TRIAL: NCT06411483
Title: Determining the Physiological Mechanisms Behind the ObeEnd Device on Factors Regulating Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Sylvia Santosa, Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 30015228
Record Dates: First submitted 2024-03-26; First posted 2024-05-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy Obesity, Metabolically; Obesity
Keywords: acupuncture; obesity; appetite; weight
MeSH Terms: conditions — Obesity, Metabolically Benign; Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: An active device arm will be compared to an inactive device (placebo) arm
Who Masked: Participant
Masking Description: Participants will be randomized to receive active or placebo (inactive) bands.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Band (Active Comparator): Participants in this group will receive an active band which provides electrostimulation at PC6
  Interventions: Device: ObeEnd Band
- Placebo (Placebo Comparator): Participants in this group will receive an inactive band which does not provide any electrostimulation when turned on.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: ObeEnd Band — The ObeEnd band provides electrostimulation to the PC6 acupuncture point on the wrist for 30 minutes.
  Arms: Active Band
Other: Placebo — The nonfunctional ObeEnd band does not provide electrostimulation to the PC6 acupuncture point on the wrist for 30 minutes.
  Arms: Placebo

SUMMARY:
In Canada, over 60% of adults are classified as overweight and obese resulting in a public health crisis including increasing health care costs and negatively impacting the well-being of many Canadians. To overcome these barriers, the ObeEnd device, manufactured by WAT Medical Enterprise, is a new and innovative wellness technology that uses electrical pulses to stimulate acupressure point PC6 to help control appetite. PC6 stimulation could potentially modulate appetite and restore gastric dysfunction, which are important factors that contribute to obesity. If PC6 electrostimulation facilitates the normalization of appetite and restoration of gastric dysfunction in those with obesity, then the device could be a potentially helpful aid to weight loss.

To measure the change of appetite hormones and enzymes related to appetite regulation after using the ObeEnd device. The investigators hypothesize that, compared to placebo, electrostimulation of PC6 an acupuncture spot on the wrist over a two-week period will result in changes in enterogastic hormones in a direction that decreases appetite. The investigators also hypothesize that these changes will not affect physical activity levels but will correspond to changes in appetite and diet. This study will provide the first evidence of the effects of electrostimulation at PC6 on factors affecting body weight regulation providing insight into the utility of the ObeEnd device for weight control.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 kg/m2
* no history of chronic illness or disease
* premenopausal

Exclusion Criteria:

* pregnant, breastfeeding
* medications that may affect outcomes
* chronic disease or conditions that may affect outcomes
* smoking or use of nicotine containing products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Factors involved with appetite regulation | after 2 weeks of wearing the band
  Blood hormones and proteins involved with appetite regulation. Appetite will be assessed via the Adult Eating Behaviour Questionnaire to see changes from baseline. This is a 35-item questionnaire that assesses 8 traits of appetite/hunger on a 1-5 Likert scale with a score of 1 indicating "strongly disagree" and a score of 5 indicating "strongly agree" to the statement.
Dietary assessment | after 2 weeks of wearing the band
  Changes in dietary intake will be measured through 3 day food records combined with photos.
Physical activity | after 2 weeks of wearing the band
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ) to see changes from baseline. The questionnaire measures various dimensions of physical activity over a 7 day retrospective period. The questions are open ended, asking participants to fill out a number for the time period being asked. For example, "___days per week".

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Santosa, PhD, RD, Principal Investigator — Concordia University, Montreal
Locations (1):
- School of Health, Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
On request and approval by ethics
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available after the study results have been accepted for publication. The data will be available for 5 y.
Access Criteria: On request with ethics approval.